CLINICAL TRIAL: NCT02686177
Title: Effect of GLP-1 on Angiogenesis, Angiosafe Type 2 Diabetes Study 1
Brief Title: Effect of GLP-1 on Angiogenesis
Acronym: ANGIOSAFE 1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P140710; 2015-002930-35 (Other: IDRCB)
Record Dates: First submitted 2016-02-15; First posted 2016-02-19 (Estimated); Last update posted 2021-06-15 (Actual); Status verified 2021-06

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes; Angiogenesis; Liraglutide; Glucagon like peptide 1 receptor agonist
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Liraglutide; Metformin; Sulfonylurea Compounds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1: Liraglutide (Experimental): Liraglutide 1,2 mg once daily subcutaneous injection for 1 month (4 weeks)
  Interventions: Drug: Liraglutide
- 2: Add on oral antidiabetic medication (Active Comparator): Metformin or sulfonylurea depending on monotherapy
  Interventions: Drug: Metformin or sulfonylurea

INTERVENTIONS:
Drug: Liraglutide
  Arms: 1: Liraglutide
Drug: Metformin or sulfonylurea
  Arms: 2: Add on oral antidiabetic medication

SUMMARY:
GLP-1 receptor agonists are introduced in the treatment of type 2 Diabetes (T2D) and their efficacy is documented. However, safety aspects are also important to evaluate with respect to micro and macrovascular complications associated with T2D. Few studies have properly addressed the role of GLP-1-based therapies in regulating vascular integrity and angiogenesis. The study evaluate the impact of one-month treatment Liraglutide on both ANGPT2 and ANGLPT4 levels and endothelial circulating progenitor cells, angiogenesis biomarkers in type 2 diabetic patients.

DETAILED DESCRIPTION:
GLP-1 receptor agonists are introduced in the treatment of type 2 Diabetes (T2D) and their efficacy is documented. Beside their therapeutic benefits, direct cardiovascular effects have also been reported. However, safety aspects are also important to evaluate with respect to micro and macrovascular complications associated with T2D. T2D patients treated with GLP-1 analogs may suffer from microvascular complications such as macular oedema and proliferative retinopathy, characterized by excessive retinal angiogenesis. Few studies have properly addressed the role of GLP-1-based therapies in regulating vascular integrity and angiogenesis. The role of GLP-1 on endothelial cell (EC) growth, EC integrity and angiogenesis thus needs to be characterized. Our aim is to provide the proof of concept that agonists of GLP-1 regulate angiogenesis in humans and identify the underlying mechanisms. The present project is the translational part of the ANR Angiosafe-T2D, regarding clinical safety aspects of GLP-1 receptor agonists (namely Liraglutide) on angiogenesis.

The study evaluate the impact of one-month treatment Liraglutide on both ANGPT2 and ANGLPT4 levels and endothelial circulating progenitor cells, angiogenesis biomarkers in type 2 diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic patients (ADA criteria)
* Age > 18 years
* Obesity (BMI >= 25 kg/m2)
* HbA1c > 6.5 %
* Treatment with Metformin and/or secretagogues
* Effective contraception (women)

Exclusion Criteria:

* Treatment with Exenatide, Liraglutide or other incretinergic regimen (<1 month before recruitment)
* Type 1 diabetes
* acute disease or infection
* chronic renal failure (MDRD eGFR≤50 mL/min)
* recent cardiovascular event or surgery (<3 months)
* pancreatitis history
* anti-VEGF treatment
* untreated cancer
* immunological disorders
* pregnancy and lactation
* Vulnerable people : deprivation of Liberty safeguards
* hypersensitivity to the active substance or to any of the excipients of the investigational drug
* diabetic ketoacidosis
* heart failure stage 3 or 4 (NYHA III-IV)
* Hepatic insufficiency
* inflammatory bowel disease and gastroparesis
* No affiliation to the social security

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-05-18 (Actual); Primary Completion 2017-08-08 (Actual); Study Completion 2021-05-28 (Actual)

PRIMARY OUTCOMES:
Difference of ANGPTL4 concentration at 4 weeks of treatment from baseline in Liraglutide and control group | At 1 month

SECONDARY OUTCOMES:
Difference of ANGPT2 concentration at 4 weeks of treatment from baseline in Liraglutide and control group | 4 weeks
  We will use commercial ANGPT2 commercial ELISA assays
Difference of endothelial circulating progenitor cells (CD34+KDR+) concentration at 4 weeks of treatment from baseline in Liraglutide and control group | 4 weeks
  Circulating progenitor cells (EPCs) will be quantified using flow cytometry before and after one month treatment GLP-1 receptor agonist or reference treatment (control group). Briefly, after erythrocyte lysis, peripheral blood will be stained with 10µL fluorescein isothiocyanate-conjugated anti-human CD34 mAb (Becton Dickinson), 10µL phycoethrin-conjugated anti-human KDR mAb (R&D Systems), and 10µL allophycocyanin-conjugated anti-CD133 mAb (Miltenyi Biotech). The frequency of CD34+ cells, CD34+ KDR+ cells before and after GLP-1R agonist or control treatment will be determined by a two-dimensional side-scatter fluorescence dot plot analysis after appropriate gating using blood samples from above-stated recruited patients
Difference of AngiomiR-126 expression at 4 weeks of treatment from baseline in Liraglutide and control group | 4 weeks
  AngiomiR-126 will be extracted from the fresh isolated cells using the miRNeasy Mini Kit (Qiagen) microRNA expression levels will be compared between type 2 diabetic subjects, before and after one-month GLP-1R agonist treatment and in the control group
Difference of Circulating soluble adhesion molecules as endothelial activation markers: ICAM-1 and VCAM-1 concentration at 4 weeks of treatment from baseline (Liraglutide versus control group) | 4 weeks
  The measurement of circulating soluble adhesion molecules as endothelial activation markers: ICAM-1 and VCAM-1 will be done with ELISA commercial assays

CONTACTS AND LOCATIONS:
Overall Officials: Bénédicte GABORIT, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Marseille
Locations (1):
- Nutrition department, pole ENDO - Assistance Publique Hôpitaux Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gaborit B, Julla JB, Besbes S, Proust M, Vincentelli C, Alos B, Ancel P, Alzaid F, Garcia R, Mailly P, Sabatier F, Righini M, Gascon P, Matonti F, Houssays M, Goumidi L, Vignaud L, Guillonneau X, Erginay A, Dupas B, Marie-Louise J, Autie M, Vidal-Trecan T, Riveline JP, Venteclef N, Massin P, Muller L, Dutour A, Gautier JF, Germain S. Glucagon-like Peptide 1 Receptor Agonists, Diabetic Retinopathy and Angiogenesis: The AngioSafe Type 2 Diabetes Study. J Clin Endocrinol Metab. 2020 Apr 1;105(4):dgz069. doi: 10.1210/clinem/dgz069. PMID 31589290